CLINICAL TRIAL: NCT05207072
Title: Prospective Observational Trial for a Cardiac Rehabilitation eHealth Application in Post-ACS Patients; Assessment of the Effects on Sustainability and Participation Level (REHAB+)
Brief Title: Mobile Tele-Monitoring Guided Cardiac Rehabilitation in Post-Acute Coronary Syndrome Patients
Acronym: REHAB+
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, AWJ van t Hof, Professor of Cardiology, MD PhD, Maastricht University
Other Study IDs: Z20210177; 210707 (Other Grant/Funding Number: The European Institute of Innovation and Technology)
Record Dates: First submitted 2021-12-24; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Rehabilitation; Acute Coronary Syndrome
Keywords: Cardiac Telerehabilitation; Acute Coronary Syndrome; Cardiac Rehabilitation
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mobile Cardiac Rehabilitation (mCR) group: The mCR programme involves a home-based programme for 12 months in which patients are supplied with a smartphone/application with a data subscription from LIVA. Through this application patients are able to measure and register physical activity, heart frequency and intensity (BORG scale) and can monitor progress. A healthcare professional (coach) also has access to a portal to monitor progress of different patients, advice on rehabilitation approach and stimulate compliance. Together with their coaches every patient makes their own rehabilitation programme. Patients will be coached for 12 months starting intensively with decreasing amounts of contacts over time.
- Traditional Cardiac Rehabilitation (CR) group: The traditional CR programme involves standard a standard CR programme over a 6-8 weeks period. Subjects receive no advice or coaching after the end of the traditional CR program.

SUMMARY:
Cardiac rehabilitation (CR) programmes are effective measures to reduce recurrent ischemic events in post-acute coronary syndrome (ACS) patients. However, participation rates in CR programmes following myocardial infarction remain low and their long-term effects are uncertain.

Home-based CR in combination with novel innovative e-Health applications could overcome barriers to accessibility and participation. Rehab+, a mobile cardiac rehabilitation (mCR) programme co-created with patients and rehabilitation centres, is designed to future-proof CR and to make CR more accessible to patients. Moreover, Rehab+ will be offered for 12 consecutive months after myocardial infarction and could therefore result in greater sustained effects.

This prospective, investigator-initiated, multicentre, matched control, observational trial intends to enroll 900 post-ACS patients. Subjects following ACS will be enrolled in the hospital if they meet all the eligibility criteria. Each subject will be able to choose between one of the 2 treatment groups, i.e. 12 months of mCR or 6-8 weeks of traditional centre-based CR. The follow-up for each subject will take 12 months for both groups.

The primary objective of this study is to assess whether mCR programme result in better sustained effects on physical, mental and social outcomes in post-ACS patients, as compared to post-ACS patients who follow the traditional CR programme.

The main hypothesis is that mCR is expected to result in greater improvement in Quality of Life at 12 months as compared to traditional CR.

DETAILED DESCRIPTION:
Subjects will be screened during hospitalisation following myocardial infarction. All eligible patients for CR will be informed about the study and requested to participate. Those fulfilling the eligibility criteria who have provided written informed consent will be allocated based upon patient preference to the mCR group with mobile tele-monitoring guidance or the control group following the regular CR programme.

Patient data will be collected at three different time points, T0 at inclusion (baseline), T1 after 3 months and T2 after 12 months. Data will be administered from the patient's (electronic) health record collected during usual care. Extra data will be administered through questionnaires.

Patients can leave the study at any time for any reason if they wish to do so without any consequences. The site investigator can decide to withdraw a patient from the study for urgent medical reasons.

In order to assess the effects on sustained physical fitness after participation in the mCR programme it was determined that an inclusion of 300 patients per group would be sufficient to examine the aim of this study.

This is based on the expected difference in increase in Quality of Life at 12 months between the mCR and matched traditional CR group with an estimated standard deviation of 7 units (Physical component score SF-36 questionnaire) in both groups. The base correlation is expected to be 0.5. Assuming 80% power and 5% two-sided significance level (alpha=0.05), the sample size (n) required to achieve a probability of 80% of detecting a difference in the QoL level between two groups, is n=268 per group.

Based on 10% withdrawal or incomplete data, the investigators aim for a group size of n= 300 per group (n=600 in total). In order to find a control group of 300 matched patients, 600 consecutive patients following regular CR will be registered. The investigators expect patients choosing for mCR versus regular CR in a ratio of 1:2. Therefore a total of 900 patients will be included in the study.

ELIGIBILITY:
During admission after myocardial infarction all eligible patients for CR will be informed about the study and requested to participate.

Inclusion Criteria

Subjects of 18 years or older who are a candidate for CR with the following criteria:

* Patients with a myocardial infarction (both STEMI and NSTEMI);
* Signed written informed consent.

Exclusion Criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Contraindication to CR;
* Mental impairment leading to inability to cooperate;
* Severe impaired ability to exercise;
* participating in a cardiac rehabilitation programme at the time of inclusion;
* Insufficient knowledge of the native language;
* Participating in CR elsewhere.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of 18 years or older following acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life measured by the SF-36 questionnaire. | At 12 months (T2) and baseline (T0)
  Short Form 36 (SF-36) quality of life scale will be used to evaluate health-related quality of life between the end of follow-up (T2) and baseline (T0). Items are grouped in 8 scaled scores exploring multiple dimensions of health (vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning, mental health).
  Scoring will be performed as recommended by the SF-36 instruction manual to create the eight scale scores. Furthermore, these subscales sum to obtain the total SF-36 score and will be summarized into two composite scores (physical and mental quality of life).

SECONDARY OUTCOMES:
Change in Quality of Life measured by the SF-36 questionnaire. | At 3 months (T1) and baseline (T0)
  Short Form 36 (SF-36) quality of life scale will be used to evaluate health-related quality of life between 3 months (T1) and baseline (T0). Items are grouped in 8 scaled scores exploring multiple dimensions of health (vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning, mental health).
  Scoring will be performed as recommended by the SF-36 instruction manual to create the eight scale scores. Furthermore, these subscales sum to obtain the total SF-36 score and will be summarized into two composite scores (physical and mental quality of life).
Rate of re-hospitalization or visits to the emergency department. | At 12 months (T2)
  The occurrence of re-hospitalizations or visits to the emergency department between baseline and the end of follow-up.
Change in physical activity as measured by the International Physical Activity Questionnaire (IPAQ). | At 12 months (T2), 3 months (T1) and baseline (T0)
  The IPAQ short form (IPAQ-sf) with an activity diary (in minutes/week) will be used to evaluate the physical activity level of the participants. Results will be reported in categories (low activity levels, moderate activity levels or high activity levels).
Self-reported impact of eHealth on its users measured by the e-Health Impact Questionnaire (eHIQ). | At 3 months (T1)
  The eHealth Impact Questionnaire (eHIQ) measures users' attitudes towards an application which they recently viewed. It is divided into the 11-item eHIQ-Part 1, asking for general attitudes towards using the internet to access health information and the 26-item eHIQ-Part 2, which is related to the effects of using a specific health-related application on three subscales: 1) confidence and identification, 2) information and presentation and 3) understanding and motivation. Both answering formats range from 1 (strongly disagree) to 5 (strongly agree). Part 1 will be assessed in both groups, while part 2 will only be assessed in the mCR group.
Change in metabolic equivalent of task (MET) as calculated from treadmill or cycle ergometry. | At 12 months (T2) and baseline (T0)
  Physical fitness level will be measured as number of MET during an incremental maximal exercise test (cycling or treadmill). The test will be performed under supervision. All tests will be performed by the same protocol. For patients who are not able to participate cycling test, this test will be replaced by the treadmill Test. The testing modality chosen per centre at T0, will remain the same at T2. To ensure a safe environment in which the tests can be performed, the test will be performed to applicable guidelines and regulations within each participating centre.
Change in lipid profile | At 12 months (T2), at 3 months (T1) and at baseline (T0)
  Blood samples as part of standard care will be obtained to assess changes in lipid profiles (in mmol/L).
Change in HbA1c | At 12 months (T2), at 3 months (T1) and at baseline (T0)
  Blood samples as part of standard care will be obtained to assess changes in HbA1c (in mmol/mol).
Change in smoking (tobacco addiction) according to the Fagerström test. | At 12 months (T2), at 3 months (T1) and at baseline (T0)
  The Fagerström test consists of six questions. The minimum value is 0 points and maximum values is 10 points. The higher score represents the greater nicotine dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Arnoud van 't Hof, MD PhD, Principal Investigator — Maastricht University
Locations (4):
- Stichting Zuyderland Medisch Centrum, Heerlen, Limburg, Netherlands
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen de la Victoria de Málaga, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Mierlo RFR, Houben VJG, Rikken SAOF, Gomez-Doblas JJ, Lozano-Torres J, van 't Hof AWJ. Cardiac (tele)rehabilitation in routine clinical practice for patients with coronary artery disease: protocol of the REHAB + trial. Front Cardiovasc Med. 2024 Jul 29;11:1387148. doi: 10.3389/fcvm.2024.1387148. eCollection 2024. PMID 39224752
- See also: Links to the REHAB+ project on the website of the grant funding organization (European Institute of Innovation and Technology). — https://eit-health.de/en/rehabplus/